CLINICAL TRIAL: NCT00278265
Title: First Line Therapy With Methotrexate (MTX) and Second Line Therapy With Fludarabine of Patients With T-Cell Large Granular Lymphocyte Leukemia (T-LGL)
Brief Title: Methotrexate Followed by Fludarabine in Patients With T-Cell Large Granular Lymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: German CLL Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LGL1; GCLLSG-LGL1; EU-20564; CDR0000454596 (Other: Clinical Data Repository)
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: T-Cell Large Granular Lymphocytic Leukemia
Keywords: T-cell large granular lymphocyte leukemia; anemia; neutropenia
MeSH Terms: conditions — Leukemia, Large Granular Lymphocytic; Anemia; Neutropenia | interventions — Methotrexate; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MTX followed by fludarabine (Experimental): MTX is given with a dose of 10-20mg weekly Fludarabine is dosed with 25mg/m2 day 1-3 of 28 days, up to 4 cycles
  Interventions: Drug: MTX followed by fludarabine

INTERVENTIONS:
Drug: MTX followed by fludarabine — MTX should be administered with 10-20mg weekly, calculated according to the body weight. Fludarabine should be administered with 25mg/m2 on day 1-3 of 28 days, up to 4 cycles
  Other Names: methotrexate, fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as methotrexate and fludarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well methotrexate works as first-line therapy and fludarabine works as second-line therapy in treating patients with T-cell large granular lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine remission rates and duration of remission in patients with T-cell large granular lymphocytic (T-LGL) leukemia needing intervention because of anemia or neutropenia and are treated with parenteral methotrexate (MTX) as first-line therapy
* Determine remission rate and duration of remission in patients who fail to respond to MTX therapy and are subsequently treated with fludarabine as second-line therapy.

Secondary

* Determine the side effects of these drugs in these patients.
* Determine the rate of molecular remissions in patients treated with these drugs.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

Patients receive methotrexate subcutaneously once weekly in the absence of disease progression or unacceptable toxicity. Patients not achieving a response to methotrexate receive fludarabine IV on days 1-3. Treatment with fludarabine repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of T-cell large granular lymphocytic (T-LGL) leukemia
* Must have concurrent anemia or neutropenia

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 2 years
* Not pregnant
* Fertile patients must use effective contraception
* No other malignancy
* No active infection

PRIOR CONCURRENT THERAPY:

* No prior immunosuppressive treatment
* No previous treatment with methotrexate or fludarabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 12 months after inclusion in the study
  he remission status was assessed according to the guidelines of the National Cancer Institute Sponsored Working Group (NCI-WG) [20 Cheson BD, Bennett JM, Grever M, et al. National Cancer Institute-sponsored Working Group guidelines for chronic lymphocytic leukemia: revised guidelines for diagnosis and treatment. Blood 1996; 87: 4990-4997.]. Restaging after the end of treatment included evaluation of the peripheral blood and physical examination; use of imaging techniques (ultrasound and conventional radiography or computertomography) and evaluation of the bone marrow were mandatory to assign a complete remission

SECONDARY OUTCOMES:
Duration of remission | up to 24 months after inclusion in the study
  he remission status was assessed according to the guidelines of the National Cancer Institute Sponsored Working Group (NCI-WG) [20 Cheson BD, Bennett JM, Grever M, et al. National Cancer Institute-sponsored Working Group guidelines for chronic lymphocytic leukemia: revised guidelines for diagnosis and treatment. Blood 1996; 87: 4990-4997.]. Restaging after the end of treatment included evaluation of the peripheral blood and physical examination; use of imaging techniques (ultrasound and conventional radiography or computertomography) and evaluation of the bone marrow were mandatory to assign a complete remission
Molecular remission rate | 2 months after the last dose of study medication
Adverse events rate and severity | up to 28 days after the last dose of study medication
  Adverse events were reported according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC version 2.0)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kneba, Study Chair — University Hospital Schleswig-Holstein
Locations (7):
- Germany (7):
  - Robert Roessle Comprehensive Cancer Center - Charite Campus Buch, Berlin
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - I. Frauenklinik und Hebammenschule der Ludwig-Maximillians Universitaet Muenchen, Munich
  - Klinikum Schwaebisch Gmuend Stauferklinik, Mutlangen
  - Praxis fuer Haematologie und Interne Onkologie, Norderstedt
  - St. Marien - Krankenhaus Siegen GMBH, Siegen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No